CLINICAL TRIAL: NCT02737748
Title: A Phase I/II Study to Evaluate the Safety and Efficacy of TWB-103 in Adult Patients With Split-Thickness Skin Graft Donor Site Wounds (DSW)
Brief Title: TWB-103 for Adult Patients With Split-Thickness Skin Graft Donor Site Wounds
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Transwell Biotech Co., Ltd. (Industry)
Collaborators: A2 Healthcare Taiwan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-FDF-C001
Record Dates: First submitted 2016-03-28; First posted 2016-04-14 (Estimated); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-06

CONDITIONS: Donor Site Complication
Keywords: Donor Site Wounds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TWB-103 Group (Experimental): Subjects will receive TWB-103 2 to 3 times till 100% re-epithelialization or up to 10 days (around once every 3 days).
  Interventions: Drug: TWB-103 Group
- Placebo Group (Placebo Comparator): Subjects will receive placebo 2 to 3 times till 100% re-epithelialization or up to 10 days (around once every 3 days).
  Interventions: Drug: Placebo Group

INTERVENTIONS:
Drug: TWB-103 Group — Each subject received TWB-103+Tegaderm for up to 10 days or to the day of 100% re-epithelialization, whichever comes first, followed by Tegaderm alone application from Day 10 to 14 if failing to achieve 100% re-epithelialization by Day 10.
  Other Names: TWB-103+Tegaderm
  Arms: TWB-103 Group
Drug: Placebo Group — Each subject received Placebo+Tegaderm for up to 10 days or to the day of 100% re-epithelialization, whichever comes first, followed by Tegaderm alone application from Day 10 to 14 if failing to achieve 100% re-epithelialization by Day 10.
  Other Names: Placebo+Tegaderm
  Arms: Placebo Group

SUMMARY:
Primary objective:

1. To evaluate the safety of TWB-103 in split-thickness skin graft donor site wounds (DSW) for Phase I in terms of Incidence of treatment-related AEs and SAEs (including infections and bleeding)
2. To evaluate the efficacy for Phase I+II of TWB-103 in split-thickness skin graft donor site wounds (DSW) in terms of The healing time from DSW creation to 100% re-epithelialization

Secondary objective:

1. To evaluate the efficacy of TWB-103 in split-thickness skin graft donor site wounds (DSW) in secondary efficacy endpoints
2. To evaluate the safety of TWB-103 in split-thickness skin graft donor site wounds (DSW) in secondary safety endpoints

DETAILED DESCRIPTION:
The study was designed to evaluate the safety and efficacy of the TWB-103 in adult subjects with split-thickness skin graft donor site wounds (DSW). In Phase I proportion, eligible subjects were recruited sequentially with one week staggering of treatment. Eligible subjects were randomized into TWB-103 or Placebo groups in a 1:1 ratio. Phase I was planned to recruit 3 evaluable subjects each in TWB-103 and Placebo groups. Evaluable subjects in Phase I were (1) he/she who received at least one dose and had follow-up evaluation at least 14 days after the first dose or (2) he/she who received at least one dose and had early withdrawn due to safety reasons before Day 28. When all of those 6 evaluable subjects completed the planned treatment period (14 days or till first 100% re-epithelialization, which came first), the recruitment was temporarily stopped for 14 days for safety observation. The safety data before and on Day 28 Visit were reviewed by the sponsor and the principal investigator. If no safety issue was decided, the study would enter Phase II portion and eligible subjects would be randomized into a 1:1 ratio into one of the TWB-103 and Placebo groups. The dosing regimen designed in Phase II portion was the same as it was designed in Phase I portion.

Subjects were instructed to attend scheduled visits at Screening, Day 0 (treatment start the day), Day 3, Day 7, Day 10, and Day 14 (end of treatment). All subjects were scheduled to attend a follow-up visit on Day 28 to evaluate the status of the target wound and then enter a 360-day follow-up phase. During the 360-day follow-up, four follow-up visits were scheduled at 90±14 days, 180±14 days, 270±14 days, and 360±14 days following the subject's Day 28 visit (if no Day 42 visit) or Day 42 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Female/male patients, aged 20-65 years old
2. Presenting a split-thickness skin graft donor site wound with a minimum size of 15 cm2 but no more than 100 cm2, with a minimum width of 3 cm and with an approximate thickness of 0.010~0.012 inches. The graft cannot be harvested from a site from which a skin graft was previously obtained.
3. If the primary wound is a result of a thermal or chemical burn, the total body surface area of the said wound must be less than 15%.
4. Females of childbearing potential must have a documented negative serum pregnancy test done at the screening visit, which is within 2 weeks prior the DSW creation and the treatment
5. Both male and female patients must agree to use highly effective contraceptives from signing informed consent to 30 days after the last dose administration.
6. Willing to comply with the study protocol and to sign the Informed Consent Form

Exclusion Criteria:

1. Female patients who are pregnant or lactating or planning a pregnancy and any male patient whose partner (wife) planning a pregnancy from signing informed consent to 30 days after the last dose administration.
2. Clinically significant disease or condition that may compromise graft take and/or donor site healing (e.g. the presence of a bleeding disorder, capillary fragility, venous or arterial disorder directly affecting the donor site to be treated, known or suspected systemic malignancies, human immunodeficiency virus infection, renal or liver disease, uncontrolled diabetes mellitus, thrombocytopenia, vasculitis, poor nutritional status).
3. Patients who are currently receiving or have received the following treatments within 4 weeks prior to study entry are excluded from the study:

   1. systemic or inhaled corticosteroids or immunosuppressant agents; or
   2. therapeutic doses of anticoagulants (e.g. Coumadin, Heparin, low molecular weight Heparin) for pre-existing medical conditions, for whom a dose interruption from Screening through the end of the study period is contraindicated.
4. Autoimmune disease, e.g. lupus erythematosus, multiple sclerosis.
5. Hematologic disease, malignancy or hypo-immunity.
6. History of HIV or congenital immunodeficiency.
7. History of alcoholism or drug abuse.
8. Have used any tobacco product within 1 week prior to Day 0.
9. Patients previously treated with any cell-based product, including autologous tissue at the treatment site.
10. Received an investigational drug, device or biological/bioactive treatment within 30 days prior to Screening Visit.
11. Any clinical condition or significant concurrent disease judged by the investigator to complicate the evaluation of the trial treatment.
12. History of sensitivity to bovine or porcine origin materials, or human serum albumin.
13. DSWs located in the face, over joints, lower legs or the buttocks
14. Any of the following hematologic abnormalities: (Hemoglobin < 10.0 g/dL, ANC < 1,500/μL, platelets < 75,000 /μL)
15. Any of the following serum chemistry abnormalities: (Total bilirubin > 1.5 × ULN, AST or ALT > 3 × ULN, gamma-GT > 2.5 x ULN, Alk-P > 2.5 x ULN, serum albumin < 2.7 g/dL, creatinine >1.5 x ULN, any other ≥ Grade 2 laboratory abnormality (based on CTCAE) at baseline (other than those listed above)
16. DSWs in area with active skin infection or with skin condition that is considered highly susceptible to infection judged by the investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niann-Tzyy Dai, MD, PhD., Principal Investigator — Tri-Service General Hospital
Locations (3):
- Japan (2):
  - Nippon Medical School, Tokyo
  - Tokyo Medical University, Tokyo
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study enrolling subjects from one site in Taiwan and two sites in Japan, between July 06, 2017 and May 07, 2021.
Pre-assignment Details: 48 subjects were screened in this study; 8 subjects were screen failures, resulting in 40 randomized subjects.
Groups:
- TWB-103 Group: Each subject received TWB-103+Tegaderm for up to 10 days or to the day of 100% re-epithelialization, whichever comes first, followed by Tegaderm alone application from Day 10 to 14 if failing to achieve 100% re-epithelialization by Day 10. For all assessments, the baseline was defined as the most recently available data before the administration of 1st dose treatment.
- Placebo Group: Each subject received Placebo+Tegaderm for up to 10 days or to the day of 100% re-epithelialization, whichever comes first, followed by Tegaderm alone application from Day 10 to 14 if failing to achieve 100% re-epithelialization by Day 10. For all assessments, the baseline was defined as the most recently available data before the administration of 1st dose treatment.
Period: Overall Study
Arm/Group | TWB-103 Group | Placebo Group
Started | 20 | 20
Phase I | 3 | 4
Phase II | 17 | 16
Completed | 19 | 18
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Groups:
- TWB-103 Group: Each subject received TWB-103+Tegaderm for up to 10 days or to the day of 100% re-epithelialization, whichever comes first, followed by Tegaderm alone application from Day 10 to 14 if failing to achieve 100% re-epithelialization by Day 10. The baseline was defined as the most recently available data before the administration of 1st dose treatment.
- Placebo Group: Each subject received Placebo+Tegaderm for up to 10 days or to the day of 100% re-epithelialization, whichever comes first, followed by Tegaderm alone application from Day 10 to 14 if failing to achieve 100% re-epithelialization by Day 10. The baseline was defined as the most recently available data before the administration of 1st dose treatment.
- Total: Total of all reporting groups
Arm/Group | TWB-103 Group | Placebo Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (14.53) | 42.2 (14.56) | 43.5 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 20 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 5 | 5 | 10
  Taiwan | 15 | 15 | 30
Baseline Donor Site Wound (DSW) Size [Mean (Standard Deviation); unit: cm^2] | 53.37 (18.726) | 40.91 (19.427) | 47.14 (19.863)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related AEs and SAEs (Including Infections and Bleeding)
Description: The number of participants with treatment-related AEs and SAEs (including infections and bleeding) will be observed for the 7 patients in Phase I
Time Frame: Day 0~Day 28
Population: Phase I was planned to recruit 3 evaluable subjects each in TWB-103 and Placebo groups. Evaluable subjects in Phase I were (1) he/she who received at least one dose and had follow-up evaluation at least 14 days after the first dose or (2) he/she who received at least one dose and had early withdrawn due to safety reasons before Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 3 | 4
Participants
  Treatment-Related AEs | 0 | 0
  SAEs | 0 | 0

2. Primary Outcome: The Healing Time From DSW Creation to the First 100% Re-epithelialization With Confirmation for at Least 10 Days Apart Assessed by the Investigator
Description: The healing time from DSW creation to the first 100% re-epithelialization with confirmation for at least 10 days apart assessed by the investigator for all patients in Phase I and II.
Time Frame: Days 42 or earlier
Population: Case first 100% re-epithelialization at any visit till Visit 7 (Day 28 Visit) with confirmation for at least 10 days apart:
  Healing Time [days] = date of first 100% re-epithelialization - date of DSW creation (Visit 2).
  Case else: Censored Healing Time [days] = date of last assessment up to Visit 7 - date of DSW creation (Visit 2).
Measure: Median (95% Confidence Interval); unit: Healing Time [days]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 19 | 14
Healing Time [days] | 9 [8.0 to 15.0] | 10 [8.0 to 15.0]
Statistical Analysis 1: Comparison: TWB-103 Group vs Placebo Group; Test type: Other; p = 0.2217, Cochran-Mantel-Haenszel

3. Primary Outcome: Number of Participants Reached Confirmed Healing Within 28 Days.
Description: The number of participants in Phase I and II reached confirmed healing by the investigator within 28 days.
Time Frame: Days 42 or earlier
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants | 19 | 14
Statistical Analysis 1: Comparison: TWB-103 Group vs Placebo Group; Test type: Other; p = 0.0324, Cochran-Mantel-Haenszel

4. Secondary Outcome: The Healing Time From DSW Creation to the First 100% Re-epithelialization With Confirmation for at Least 10 Days Apart, Assessed by the First Additional Evaluator
Description: The healing time from DSW creation to the first 100% re-epithelialization with confirmation for at least 10 days apart assessed by the investigator for all patients in Phase I and II. The first additional evaluator judged the healing status by looking at the photos of DSW.
Time Frame: Days 42 or earlier
Population: The additional evaluator who was not aware of the treatment groups would assess the wound based on the photos.
  Case first 100% re-epithelialization at any visit till Visit 7 (Day 28 Visit) with confirmation for at least 10 days apart:
  Healing Time [days] = date of first 100% re-epithelialization - date of DSW creation (Visit 2).
  Case else: Censored Healing Time [days] = date of last assessment up to Visit 7 - date of DSW creation (Visit 2).
Measure: Mean (Standard Error); unit: Healing Time [days]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 10 | 7
Healing Time [days] | 20 (2.2) | 13 (0.7)
Statistical Analysis 1: Comparison: TWB-103 Group vs Placebo Group; Test type: Other; p = 0.3975, Log Rank

5. Secondary Outcome: Number of Participants With Complete Wound Closure at Day 7, 10 and 14 After DSW Creation.
Description: Complete wound closure is defined as skin 100% re-epithelialization without drainage or dressing requirements. This endpoint will be in all patients in Phase I and II.
Time Frame: Day 7, 10 and 14
Population: Healing rates (complete wound closure) of subjects at Days 7, 10, and 14 after DSW creation were analyzed. Due to the study design, subjects would skip the following treatment visits when their wound was completely closed, resulting in the smaller subject numbers at Visit 5 (N=18) and Visit 6 (N=10). To rectify this issue, post-hoc LOCF analysis was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  Adjusted Visit 4 (Day 7) with LOCF | 9 | 11
  Adjusted Visit 5 (Day 10) with LOCF | 15 | 15
  Adjusted Visit 6 (Day 14) with LOCF | 18 | 18

6. Secondary Outcome: The Healing Percentage of Wounds (Ratio of Healing Area and Original Area) at Days 7, 10 and 14 After DSW Creation
Description: The healing percentage of wounds will be calculated based on the healing area measured on Day 7, 10 and 14, comparing to the original area measured on Day 0 for all patients in Phase I and II.
Time Frame: Day 7, 10 and 14
Population: Healing percentage was measured by the study investigator. Due to the study design, subjects would skip the following treatment visits when their wound was completely closed, resulting in the smaller subject numbers at Visit 5 (N=18) and Visit 6 (N=10). To rectify this issue, post-hoc LOCF analysis was performed.
Measure: Least Squares Mean (Standard Error); unit: Healing Percentage (%)
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Healing Percentage (%)
  Adjusted Visit 4 (Day 7) with LOCF | 65.36 (8.676) | 62.60 (8.676)
  Adjusted Visit 5 (Day 10) with LOCF | 89.20 (5.111) | 83.74 (5.111)
  Adjusted Visit 6 (Day 14) with LOCF | 88.56 (5.159) | 83.51 (5.159)

7. Secondary Outcome: The Pain Change From Baseline to Post-wound Creation Visits Based on Short-form McGill Pain Questionnaire Score
Description: All patients in Phase I and II will evaluate the pain based on Short-form McGill pain questionnaire at each visit.
  The visual analogue scale (VAS) for pain is a continuous scale comprised of a horizontal line, usually, 10 cm (= 100 mm) in length, scored from 0 (none) to 10 (extreme). On this scale, a higher score in VAS indicates the worse pain.
Time Frame: Days 3, 7, 10, 14, 28, 42, Day 90/180/270/360 from Day 28 or 42
Population: The pain assessment was measured by employing short-form McGill pain questionnaire at all scheduled visits, except Visit 2 (Day 0). The visual analogue scale (VAS) for pain is a continuous scale comprised of a horizontal line, usually, 10 cm (= 100 mm) in length, scored from 0 (none) to 10 (extreme). On this scale, a higher score in VAS indicates the worse pain.
Measure: Mean (Standard Deviation); unit: VAS (0~10 cm)
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
VAS (0~10 cm)
  Baseline | 1.89 (2.833) | 1.06 (2.399)
  Adjusted Visit 3 (Day 3) | 1.79 (2.137) | 1.58 (2.091)
  Adjusted Visit 4 (Day 7) | 0.82 (1.313) | 0.40 (0.701)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 0.80 (0.763) | 1.02 (1.731)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 0.38 (0.522) | 1.48 (2.062)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 20 | 19
  Adjusted Visit 7 (Day 28) | 0.37 (0.713) | 0.35 (0.943)
  Adjusted Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Adjusted Visit 8 (Day 42) | 0.45 (0.636) | 0.00 (0.000)
  Visit 9 (FU 3 Months): number analyzed (Participants) | 20 | 18
  Visit 9 (FU 3 Months) | 0.40 (1.588) | 0.06 (0.236)
  Visit 10 (FU 6 Months): number analyzed (Participants) | 19 | 18
  Visit 10 (FU 6 Months) | 0.00 (0.000) | 0.000 (0.000)
  Visit 11 (FU 9 Months): number analyzed (Participants) | 18 | 18
  Visit 11 (FU 9 Months) | 0.05 (0.212) | 0.00 (0.00)
  Visit 12 (FU 12 Months): number analyzed (Participants) | 19 | 18
  Visit 12 (FU 12 Months) | 0.04 (0.161) | 0.00 (0.00)

8. Secondary Outcome: Number of Participants With AEs and SAEs
Description: The number of participants with AEs and SAEs will be analyzed for all patients in Phase I and II.
Time Frame: Screening~ Day 360 from Day 28 or 42
Population: 40 subjects (20 in TWB-103 group and 20 in Placebo group) were included in the population for safety analysis. Treatment-emergent adverse events (TEAE) were classified as treatment-related AE, Grade 3 or greater AE, AE that required to take special actions, SAE, or SUSAR during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  AE | 7 | 10
  Treatment-Related AE | 0 | 0
  Grade≥3 AE | 0 | 0
  Grade ≥ 3 Treatment-Related AE | 0 | 0
  AE Leading to Action Taken | 0 | 0
  AE Leading to Drug withdrawn | 0 | 0
  SAE | 0 | 0
  Death SAE | 0 | 0
  SUSAR | 0 | 0
  Death SUSAR | 0 | 0

9. Secondary Outcome: Changes in Post-treatment Physical Examination Compared to Baseline
Description: Changes in post-treatment physical examination will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The physical examination of each subject was examined at all scheduled visits.
Measure: Number; unit: Participant with Physical Abnormality
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participant with Physical Abnormality
  Adjusted Visit 3 (Day 3) (Multi-Selection by Body System) | 1 | 0
  Adjusted Visit 4 (Day 7) (Multi-Selection by Body System) | 1 | 0
  Adjusted Visit 5 (Day 10) (Multi-Selection by Body System): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) (Multi-Selection by Body System) | 0 | 0
  Adjusted Visit 6 (Day 14) (Multi-Selection by Body System): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) (Multi-Selection by Body System) | 0 | 0
  Adjusted Visit 7 (Day 28) (Multi-Selection by Body System): number analyzed (Participants) | 20 | 19
  Adjusted Visit 7 (Day 28) (Multi-Selection by Body System) | 1 | 0
  Visit 8 (Day 42) (Multi-Selection by Body System): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) (Multi-Selection by Body System) | 0 | 0

10. Secondary Outcome: Changes in Post-treatment Vital Signs-pulse Rate Compared to Baseline
Description: Changes in post-treatment vital signs-pulse rate will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The vital signs-pulse rate of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Pulse Rate [beats/min]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Pulse Rate [beats/min]
  Baseline | 71.95 (10.359) | 73.90 (15.001)
  Adjusted Visit 3 (Day 3) | 74.25 (11.964) | 78.20 (13.332)
  Adjusted Visit 4 (Day 7) | 74.70 (9.314) | 73.55 (11.821)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 77.67 (11.554) | 72.33 (8.732)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 84.20 (17.021) | 82.40 (7.092)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 20 | 19
  Adjusted Visit 7 (Day 28) | 75.15 (12.119) | 74.79 (12.376)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 71.00 (2.828) | 76.00 (2.828)

11. Secondary Outcome: Changes in Post-treatment Vital Signs-body Temperature Compared to Baseline
Description: Changes in post-treatment vital signs-body temperature will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The vital signs-body temperature of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Body Temperature [degree C]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Body Temperature [degree C]
  Baseline | 36.29 (0.315) | 36.21 (0.415)
  Adjusted Visit 3 (Day 3) | 36.54 (0.463) | 36.33 (0.412)
  Adjusted Visit 4 (Day 7) | 36.47 (0.455) | 36.52 (0.465)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 36.72 (0.529) | 36.29 (0.289)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 36.44 (0.358) | 36.36 (0.207)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 20 | 19
  Adjusted Visit 7 (Day 28) | 36.35 (0.363) | 36.33 (0.333)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 36.30 (0.141) | 36.35 (0.212)

12. Secondary Outcome: Changes in Post-treatment Vital Signs-systolic Blood Pressure Compared to Baseline
Description: Changes in post-treatment vital signs-systolic blood pressure will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The vital signs-systolic blood pressure of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Systolic Blood Pressure [mmHg]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Systolic Blood Pressure [mmHg]
  Baseline | 116.80 (17.665) | 116.65 (15.792)
  Adjusted Visit 3 (Day 3) | 123.45 (16.794) | 120.30 (21.293)
  Adjusted Visit 4 (Day 7) | 118.85 (12.783) | 121.95 (15.278)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 117.44 (13.436) | 117.11 (15.584)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 119.80 (17.584) | 120.00 (13.304)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 20 | 19
  Adjusted Visit 7 (Day 28) | 124.60 (10.928) | 121.21 (11.622)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 140.00 (12.728) | 122.00 (5.657)

13. Secondary Outcome: Changes in Post-treatment Vital Signs-diastolic Blood Pressure Compared to Baseline
Description: Changes in post-treatment vital signs-diastolic blood pressure will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The vital signs-diastolic blood pressure of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Diastolic Blood Pressure [mmHg]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Diastolic Blood Pressure [mmHg]
  Baseline | 71.25 (13.325) | 69.90 (9.910)
  Adjusted Visit 3 (Day 3) | 71.50 (12.705) | 69.15 (10.282)
  Adjusted Visit 4 (Day 7) | 69.10 (6.439) | 76.15 (13.374)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 68.22 (11.745) | 70.00 (13.739)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 77.60 (7.893) | 78.40 (11.014)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 20 | 19
  Adjusted Visit 7 (Day 28) | 71.35 (11.820) | 77.95 (13.323)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 89.50 (24.749) | 95.00 (2.828)

14. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-hematology-white Blood Cells Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-hematology-white blood cells will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-hematology-white blood cells of each subject were examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: 10^9 cells /L
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
10^9 cells /L
  Baseline | 7.93 (2.107) | 7.40 (1.785)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 7.00 (1.840) | 7.44 (2.064)
  Adjusted Visit 4 (Day 7) | 7.20 (1.638) | 7.26 (2.835)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 6.27 (0.877) | 7.19 (1.425)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 9.27 (4.634) | 7.30 (0.780)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 6.52 (2.110) | 6.99 (1.760)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 4.63 (1.025) | 6.63 (1.605)

15. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-hematology-neutrophils Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-hematology-neutrophils will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-hematology-neutrophils of each subject were examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: 10^9 cells /L
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
10^9 cells /L
  Baseline | 5.36 (1.950) | 4.65 (1.542)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 4.61 (1.604) | 4.71 (1.577)
  Adjusted Visit 4 (Day 7): number analyzed (Participants) | 19 | 20
  Adjusted Visit 4 (Day 7) | 4.54 (1.431) | 4.37 (2.322)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 8
  Adjusted Visit 5 (Day 10) | 3.93 (0.808) | 4.06 (0.747)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 6.62 (4.944) | 4.71 (0.523)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 3.94 (1.733) | 4.19 (1.128)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 2.17 (0.826) | 3.44 (0.074)

16. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-hematology-Hemoglobin Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-hematology-hemoglobin will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-hematology-hemoglobin of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Hemoglobin [g/dL]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Hemoglobin [g/dL]
  Baseline | 13.47 (1.436) | 13.84 (1.741)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 13.28 (1.981) | 13.79 (2.220)
  Adjusted Visit 4 (Day 7) | 13.38 (2.033) | 13.69 (2.002)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 12.72 (1.796) | 13.56 (1.890)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 13.22 (2.565) | 13.82 (2.572)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 13.35 (1.726) | 13.73 (1.665)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 14.05 (1.344) | 13.30 (1.697)

17. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-hematology-Hematocrit Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-hematology-hematocrit will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-hematology-hematocrit of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Hematocrit [%]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Hematocrit [%]
  Baseline | 40.60 (3.886) | 42.00 (4.920)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 40.01 (5.410) | 41.57 (6.565)
  Adjusted Visit 4 (Day 7) | 40.35 (5.706) | 41.34 (5.591)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 38.07 (4.537) | 40.07 (5.525)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 39.84 (6.529) | 40.80 (7.005)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 40.43 (4.206) | 41.33 (4.312)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 41.45 (1.768) | 42.05 (2.192)

18. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-hematology-platelets Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-hematology-platelets will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-hematology-platelets of each subject were examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
10^9 platelets/L
  Baseline | 298.95 (69.549) | 284.60 (63.444)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 290.95 (63.692) | 278.70 (79.961)
  Adjusted Visit 4 (Day 7) | 308.50 (50.055) | 279.10 (67.043)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 311.44 (67.930) | 247.22 (51.575)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 314.80 (81.174) | 225.60 (26.885)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 268.42 (68.664) | 260.11 (50.326)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 248.50 (88.388) | 290.50 (19.092)

19. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-hematology-red Blood Cells Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-hematology-red blood cells will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-hematology-red blood cells of each subject were examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
10^12 cells/L
  Baseline | 4.61 (0.558) | 4.86 (0.674)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 4.54 (0.729) | 4.82 (0.824)
  Adjusted Visit 4 (Day 7) | 4.59 (0.763) | 4.83 (0.811)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 4.19 (0.476) | 4.58 (0.892)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 4.30 (0.842) | 4.48 (0.832)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 4.60 (0.586) | 4.83 (0.639)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 4.41 (0.198) | 5.21 (0.488)

20. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-biochemistry-aspartate Aminotransferase Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-biochemistry-aspartate aminotransferase will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-biochemistry-aspartate aminotransferase of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Aspartate Aminotransferase [U/L]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Aspartate Aminotransferase [U/L]
  Baseline | 22.55 (10.773) | 21.85 (8.177)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 33.37 (46.940) | 20.00 (5.648)
  Adjusted Visit 4 (Day 7) | 24.75 (15.210) | 24.40 (9.762)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 26.44 (16.883) | 21.33 (6.837)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 45.00 (43.052) | 22.40 (12.876)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 19.05 (6.060) | 22.00 (8.931)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 32.50 (23.335) | 19.50 (3.536)

21. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-biochemistry-alanine Aminotransferase Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-biochemistry-alanine aminotransferase will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-biochemistry-alanine aminotransferase of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Alanine Aminotransferase [U/L]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Alanine Aminotransferase [U/L]
  Baseline | 25.30 (18.374) | 28.20 (16.776)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 32.79 (42.926) | 22.95 (14.125)
  Adjusted Visit 4 (Day 7) | 29.25 (24.512) | 27.15 (15.301)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 31.89 (29.570) | 26.22 (15.619)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 62.20 (54.509) | 25.20 (23.868)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 21.63 (16.780) | 28.28 (24.826)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 54.50 (62.933) | 28.00 (2.828)

22. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-biochemistry-serum Creatinine Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-biochemistry-serum creatinine will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-biochemistry-serum creatinine of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Serum Creatinine [umol/L]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Serum Creatinine [umol/L]
  Baseline | 62.68 (14.386) | 62.01 (17.022)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 58.39 (14.422) | 61.75 (18.310)
  Adjusted Visit 4 (Day 7) | 60.51 (15.129) | 63.78 (19.811)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 54.42 (17.045) | 60.21 (17.133)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 57.64 (19.016) | 63.12 (37.742)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 62.44 (12.363) | 64.63 (18.637)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 56.58 (5.001) | 66.30 (6.251)

23. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-biochemistry-blood Urea Nitrogen Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-biochemistry-blood urea nitrogen will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-biochemistry-blood urea nitrogen of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Blood Urea Nitrogen [mg/dL]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Blood Urea Nitrogen [mg/dL]
  Baseline | 13.59 (4.838) | 14.06 (4.271)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 11.58 (2.234) | 13.23 (3.779)
  Adjusted Visit 4 (Day 7): number analyzed (Participants) | 19 | 20
  Adjusted Visit 4 (Day 7) | 14.46 (3.956) | 14.72 (5.427)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 13.02 (3.938) | 13.54 (2.967)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 14.12 (5.304) | 14.48 (3.189)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 12.82 (3.873) | 13.13 (2.537)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 11.90 (2.970) | 16.50 (3.536)

24. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-biochemistry-Albumin Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-biochemistry-albumin will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-biochemistry-albumin of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Albumin [g/dL]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Albumin [g/dL]
  Baseline | 4.24 (0.411) | 4.08 (0.492)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 3.99 (0.540) | 3.87 (0.526)
  Adjusted Visit 4 (Day 7) | 4.12 (0.586) | 4.09 (0.528)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 3.86 (0.529) | 3.98 (0.377)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 4.02 (0.585) | 4.30 (0.200)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 4.31 (0.401) | 4.33 (0.387)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 4.45 (0.212) | 4.50 (0.283)

25. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-biochemistry-bilirubin Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-biochemistry-bilirubin will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-biochemistry-bilirubin of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Bilirubin [umol/L]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Bilirubin [umol/L]
  Baseline | 9.63 (4.824) | 8.10 (4.975)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 7.44 (3.842) | 8.92 (6.039)
  Adjusted Visit 4 (Day 7) | 8.39 (5.095) | 8.73 (4.876)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 9.20 (5.590) | 9.64 (4.470)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 14.30 (10.487) | 9.03 (3.058)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 9.40 (6.565) | 9.10 (2.873)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 18.22 (8.829) | 6.84 (2.419)

26. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-biochemistry-gamma-glutamyl Transferase Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-biochemistry-gamma-glutamyl transferase will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-biochemistry-gamma-glutamyl transferase of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Gamma-Glutamyl Transferase [U/L]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Gamma-Glutamyl Transferase [U/L]
  Baseline | 37.65 (36.863) | 38.75 (26.754)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 37.16 (31.597) | 37.25 (26.479)
  Adjusted Visit 4 (Day 7) | 37.60 (29.674) | 39.65 (30.275)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 44.11 (33.572) | 49.44 (39.170)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 56.20 (36.072) | 47.80 (43.200)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 28.47 (19.234) | 38.22 (33.676)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 32.50 (24.749) | 21.50 (0.707)

27. Secondary Outcome: Changes in Post-treatment General Laboratory Assessment-biochemistry-alkaline Phosphatase Compared to Baseline
Description: Changes in post-treatment general laboratory assessment-biochemistry-alkaline phosphatase will be analyzed for all patients in Phase I and II.
Time Frame: Days 3, 7, 10, 14, 28, 42
Population: The general laboratory assessment-biochemistry-alkaline phosphatase of each subject was examined at all scheduled visits.
Measure: Mean (Standard Deviation); unit: Alkaline Phosphatase [U/L]
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Alkaline Phosphatase [U/L]
  Baseline | 102.65 (74.944) | 107.65 (79.693)
  Adjusted Visit 3 (Day 3): number analyzed (Participants) | 19 | 20
  Adjusted Visit 3 (Day 3) | 97.95 (63.847) | 101.35 (73.382)
  Adjusted Visit 4 (Day 7): number analyzed (Participants) | 19 | 20
  Adjusted Visit 4 (Day 7) | 104.63 (70.811) | 102.85 (71.589)
  Adjusted Visit 5 (Day 10): number analyzed (Participants) | 9 | 9
  Adjusted Visit 5 (Day 10) | 156.22 (74.933) | 158.89 (79.899)
  Adjusted Visit 6 (Day 14): number analyzed (Participants) | 5 | 5
  Adjusted Visit 6 (Day 14) | 138.80 (101.935) | 196.40 (91.694)
  Adjusted Visit 7 (Day 28): number analyzed (Participants) | 19 | 18
  Adjusted Visit 7 (Day 28) | 108.16 (84.534) | 114.00 (82.523)
  Visit 8 (Day 42): number analyzed (Participants) | 2 | 2
  Visit 8 (Day 42) | 156.50 (118.087) | 73.50 (7.778)

28. Secondary Outcome: Number of Participants With Treatment-related AEs and SAEs (Including Infections and Bleeding)
Description: The number of participants with treatment-related AEs and SAEs (including infections and bleeding) will be observed for all patients in Phase I and II
Time Frame: Screening~ Day 360 from Day 28 or 42
Measure: Count of Participants; unit: Participants
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  Treatment-Related AEs | 0 | 0
  SAEs | 0 | 0

29. Secondary Outcome: The Number of Censored Subjects Assessed by the Investigator and the First Additional Evaluator
Description: The number of censored subjects in Phase I and II assessed by the investigator and the first additional evaluator. The first additional evaluator judged the healing status by looking at the photos of DSW. If the 100% re-epithelialization was not observed by Day 28 visit, the healing time was censored on the day of the last visit up to Day 28 visit. If the 100% re-epithelialization was observed by Day 28 visit but no confirmation was made, the healing time was censored on day of the last visit up to Day 28 visit.
Time Frame: Days 42 or earlier
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | TWB-103 Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  Investigator | 1 | 6
  First Additional Evaluator | 10 | 13

ADVERSE EVENTS:
Time Frame: Screening ~ Day 360 from Day 28 or 42
Description: The primary safety endpoint of Phase I part was the incidence of treatment-related AEs and SAEs. Among 7 subjects (3 in TWB-103 group and 4 in Placebo group) included for the evaluation. For the whole study, 40 subjects (20 in TWB-103 group and 20 in Placebo group) were included for safety analysis.
Groups:
- TWB-103 add-on Tegaderm: TWB-103 is the primary therapeutics with the use of Tegaderm as a wound-site protection
- Placebo+Tegaderm: Placebo to TWB-103 with the use of Tegaderm as a wound-site protection
Arm/Group | TWB-103 add-on Tegaderm | Placebo+Tegaderm
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 10/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TWB-103 add-on Tegaderm (N=20) | Placebo+Tegaderm (N=20)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Application site dermatitis (General disorders) | 1 (1) | 1 (1)
Application site discharge (General disorders) | 0 (0) | 2 (2)
Application site erosion (General disorders) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 2 (3) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Application site folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Some cases that healing observed by 1st evaluator could not be confirmed due to the lack of following visits. These are considered as flaws of protocol design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT02737748/Prot_SAP_000.pdf